CLINICAL TRIAL: NCT07394114
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled , Phase 3 Study Comparing the Efficacy and Safety of HDM1005 Versus Placebo in Subjects With T2DM Inadequate Glycemic Control With Diet and Exercise Alone
Brief Title: A Study of HDM1005 in Participants With Type 2 Diabetes Not Controlled With Diet and Exercise Alone
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HDM1005-302
Record Dates: First submitted 2026-02-02; First posted 2026-02-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HDM1005 1 (Experimental): HDM1005 administered subcutaneously (SC).
  Interventions: Drug: HDM1005 1
- HDM1005 2 (Experimental): HDM1005 administered SC.
  Interventions: Drug: HDM1005 2
- Placebo (Placebo Comparator): administered SC.
  Interventions: Drug: HDM1005 injection or placebo

INTERVENTIONS:
Drug: HDM1005 1 — administered SC, QW, 52 weeks.
  Arms: HDM1005 1
Drug: HDM1005 2 — administered SC, QW, 52 weeks.
  Arms: HDM1005 2
Drug: HDM1005 injection or placebo — administered SC, QW, 52 weeks.
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled , phase 3 clinical trial aimed at evaluating the efficacy and safety of HDM1005 versus placebo in subjects with T2DM inadequate glycemic control with diet and exercise alone.

A total of 240 subjects will be enrolled. All subjects will be stratified by baseline HbA1c levels (≤8.5% or >8.5%) , then randomized 1:1:1 to: Group 1 (HDM1005), Group 2 (HDM1005), and Group 3 (placebo), with 80 subjects in each treatment group. At week 36, subjects in placebo group will receive HDM1005 injection until week 52. All treatment groups will implement dose titration to achieve the target dose.

The study consists of: up to 2-week screening, 2-week run-in, 36-week core treatment, 16-week extension treatment, and 4-week follow-up, totaling 60 weeks. The end-of-study visit will be conducted 28 days after the last administration cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed as Type 2 Diabetes Mellitus (T2DM) for at least 12 weeks and have not used any antihyperglycemic medications during for at least 12 weeks prior to screening.
2. Hemoglobin A1c (HbA1c) ≥7.5% and ≤10.5% at screening; and ≥7.0% and ≤10.5% at randomization.
3. Body Mass Index (BMI) ≥22.5 kg/m2.

Exclusion Criteria:

1. Other types of diabetes besides T2DM.
2. Acute complications of diabetes (such as diabetic ketoacidosis, diabetic lactic acidosis, or hyperosmolar non-ketoticcoma) occurred within 24 weeks prior to signing the Informed Consent Form (ICF).
3. History of a level 3 hypoglycemic episode or a history of asymptomatic hypoglycemic episodes within 24 weeks prior to signing the ICF.
4. History or family history of medullary thyroid carcinoma (MTC), thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2).
5. History of acute or chronic pancreatitis; or presence of risk factors for pancreatitis; or history of symptomatic gallbladder disease requiring treatment per investigator's assessment within 24 weeks prior to signing the ICF.
6. Investigator determines that the subject has a condition or disease affecting gastric emptying or gastrointestinal nutrient absorption, such as weight-loss surgery or other gastric resections, irritable bowel syndrome, dyspepsia, or gastroparesis.
7. Use of any antidiabetic medications within 12 weeks prior to signing the ICF; excluding short-term insulin use (cumulative duration ≤7 days) for concomitant illness, stress, or perioperative periods.
8. Hemoglobin (Hb) <100 g/L (female) or <110 g/L (male).
9. FPG ≥13.9 mmol/L.
10. Aspartate aminotransferase (AST) >3× upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3× ULN.
11. Total bilirubin >1.5× ULN.
12. Fasting triglyceride (TG) >5.6 mmol/L (500 mg/dL).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-08-28 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 36
  HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline, Week 52
The percentage of patients reaching the HbA1c targets of <7.0%, ≤6.5%, and <5.7% | Week 36, Week 52
Change from baseline in fasting plasma glucose (FPG) | Baseline, Week 36, Week 52
Change from baseline in body weight | Baseline, Week 36, Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China